CLINICAL TRIAL: NCT00034606
Title: Comparing 3 Schedules of Alimta Plus Gemzar
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5115; H3E-MC-JMEL
Record Dates: First submitted 2002-05-01; First posted 2002-05-02 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasms
Keywords: Lung cancer; cancer; neoplasm; non-small; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasms | interventions — Pemetrexed; Gemcitabine

INTERVENTIONS:
Drug: Pemetrexed (Alimta) in combination with gemcitabine (Gemzar)

SUMMARY:
The purpose of the study is to measure tumor response rates for three schedules of Alimta(LY231514) in combination with gemcitabine in patients with locally advanced or metastatic non small cell lung cancer who have received no prior chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-small lung cancer
* No prior chemotherapy
* Able to care for self

Exclusion Criteria:

* An ongoing infection
* Pregnancy or breast feeding
* Other serious medical condition
* Cancer that has spread to the brain
* Inability to take folic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Rochester, Minnesota, United States